CLINICAL TRIAL: NCT06187012
Title: Hypertension Explored in Long-term Postpartum Follow-up in Later Life (HELPFUL)
Brief Title: Hypertension Explored in Long-term Postpartum Follow-up in Later Life
Acronym: HELPFUL
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 22/LO/0781
Record Dates: First submitted 2023-11-29; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Hypertension; Cardiovascular Diseases; Cerebrovascular Disorders; Vascular Diseases
Keywords: Hypertensive pregnancy; Older adults; Pre-eclampsia; Gestational hypertension; Cardiovascular risk; Disease progression; Longitudinal
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Cerebrovascular Disorders; Vascular Diseases; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 40 Years
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensive pregnancy
  Interventions: Other: Hypertensive pregnancy

INTERVENTIONS:
Other: Hypertensive pregnancy — Participants will attend one visit lasting approximately 3-4 hours on a single day or split over multiple visits to complete all measures. Participants will first be asked to provide written informed consent for the study. Participants' anthropometric measures (waist-to-hip ratio, height and weight, hip and waist circumference and left arm circumference and resting blood pressures will then be taken. After this, the participants will undergo cardiopulmonary exercise testing, followed by magnetic resonance imaging, echocardiography, retinal imaging and vascular imaging of the ear. The study visit will conclude with participants being provided with a wrist-worn physical activity monitor to wear for 7-9 days following the visit. These monitors will provide objective measures of physical activity while people go about their normal activities.

SUMMARY:
The purpose of this study is to understand more about why women who have had hypertensive pregnancies may be at increased risk of high blood pressure and why these women are often at increased risk of heart and blood vessel disease later in life.

DETAILED DESCRIPTION:
Women who experience high blood pressure during pregnancy are at increased risk of developing cardiac and vascular diseases later in life. They show changes in their heart, brain, and blood vessels long before they develop high blood pressure. The investigators therefore think that these changes develop slowly over the course of the life of the woman and establish their risk of later disease.

Through better understanding of the pattern of changes across multiple parts of the body over extended periods of time, the investigators aim to identify how advanced the underlying disease is for an individual and how the disease is likely to develop over the next few years. By comparing the rate of change across different parts of the body, the investigators can examine how one area affects another.

Data including images of the heart, brain and blood vessels will be acquired in women 10 to 25 years after their pregnancy. The initial analysis will focus on assessing differences between women who have had a normotensive pregnancy and those who have had a hypertensive pregnancy, both at a single timepoint and in changes within individuals over time.

This dataset will then be used in conjunction with previously acquired data in women who have experienced a hypertensive pregnancy to find out how patterns emerge across the whole body. The investigators will subsequently combine information from different measures at the same time and use the machine learning models to learn the patterns of change that occur as a person progresses from a healthy to a diseased state.

This will allow the researchers to identify patterns of hypertensive disease development and it may open doors to better interventions and therapies tailored towards individuals.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Participant is willing and able to give informed consent for participation in the study
  * Female who had a pregnancy 10 to 25 years prior
  * Able (in the investigator's opinion) and willing to comply with all study requirements.
  * Adequate understanding of verbal and written English

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

  * Over 10 weeks pregnant during the course of the study
  * Evidence of congenital heart disease or significant chronic disease relevant to cardiovascular or metabolic status
  * Any significant disease or disorder which, in the opinion of the investigator, might influence the participant's ability to participate in the study

For exclusion of MRI component only:

• Unsuitable for MRI based on the responses to the MRI screening form. The participant may still be included in other parts of the study.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only.
Study Population: The investigators will study a group of 200 women at 10 to 25 years postpartum to extend data coverage over time and to ensure a broad representation of hypertensive disease state during mid-life in women. This will be achieved by a follow-up of participants from a previous study called Preeclampsia Vascular Study (PVS) (08/H0604/127). These women were originally seen at 5 to 15 years post-index hypertensive or normotensive pregnancy. If required, the investigators will restart their identification and recruitment methods, previously used in PVS, based on obstetric records to identify, and recruit additional women who had pregnancies 10 to 25 years prior, to ensure that the sample size is reached. All participants will undergo a standardised imaging protocol as described in the general overview.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2042-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac right ventricular mass | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy. Index pregnancy is defined as the pregnancy which we first collected data from.
  Magnetic resonance imaging assessment of cardiac right ventricular mass indexed to body surface area (g/m^2).

SECONDARY OUTCOMES:
Cardiac left ventricular mass | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of cardiac left ventricular mass indexed to body surface area (g/m^2).
Cardiac right ventricular end-diastolic volume | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of cardiac right ventricular end-diastolic volume indexed to body surface area (ml/m^2)
Cardiac right ventricular stroke volume. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of cardiac right ventricular stroke volume indexed to body surface area (ml/m^2).
Cardiac left-ventricular end-diastolic volume. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of cardiac left ventricular end-diastolic volume indexed to body surface area (ml/m^2).
Cardiac left ventricular stroke volume | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of cardiac left ventricular stroke volume indexed to body surface area (ml/m^2).
Cardiac right ventricular systolic function | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Echocardiography assessment of right ventricular systolic function: tricuspid annular plane systolic excursion (cm).
Cardiac right ventricular ejection fraction | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of right ventricular ejection fraction measured by cardiac magnetic resonance imaging (%).
Cardiac left ventricular systolic function | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Echocardiography assessment of left ventricular systolic function
Cardiac left ventricular ejection fraction | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of left ventricular ejection fraction (%).
Cardiac right ventricular diastolic function | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Echocardiography assessment of right ventricular doppler early/late diastolic tricuspid inflow velocity ratio (E/A)
Cardiac left ventricular diastolic function | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Echocardiography assessment of left ventricular doppler early/late diastolic mitral inflow velocity ratio (E/A).
Cardiac left ventricular diastolic function | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Echocardiography assessment of left ventricular early doppler inflow velocity/peak early diastolic tissue velocity rate (E/e').
Morphology of the right ventricles | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of the right ventricles morphology using cardiac statistical atlas and principal component analysis.
Morphology of the left ventricles | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of the left ventricles morphology using cardiac statistical atlas and principal component analysis.
Aortic distensibility | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Aortic distensibility by magnetic resonance imaging (10^-3 mmHg-1).
Aortic compliance | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Aortic/central blood pressure by cuff measurement (mmHg).
Intra-hepatic liquid content and steatohepatitis | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of the liver to quantify proton density fat fraction (%).
Hepatic fibrosis | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of the liver to quantify fibro-inflammatory status from iron corrected T1 (cT1 in ms)
Renal volumes | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of renal volumes (ml/m^2).
Renal fibro-inflammatory status | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of fibro-inflammatory status from T1 (ms)
Renal blood perfusion | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Magnetic resonance imaging assessment of surrogate measures of blood perfusion from T2* (in ms).
Oxygen uptake across submaximal exercise | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Cardiopulmonary exercise test to measure oxygen uptake (ml/kg/min).
Carbon dioxide exchange kinetics across submaximal exercise | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Cardiopulmonary exercise test to measure respiratory exchange ratio (RER) calculated as carbon dioxide production divided by oxygen consumption.
Retinal arteriolar structure | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Central retinal arteriolar equivalent (CRAE) in micrometres measured using retinal imaging.
Retinal venular structure | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Central retinal venular equivalent (micrometres) measured using retinal imaging.
Retinal arteriolar-to venule diameter ratio (AVR) | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The ratio of average retinal arteriolar diameter and average retinal venous diameter (micrometres).
Ear microvascular structure. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Superior crus of anti-helix earlobe vascular calibre (micrometres) measured using ear vascular imaging.
Lung function | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The ratio of FEV1 to FVC (FEV1/FVC) measured using spirometry.
Lung capacity | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The forced vital capacity (FVC in L) measured using spirometry.
Lung volume | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The forced expiratory volume in one second (FEV1 in L) measured using spirometry.
Objective measure of vigorous physical activity. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The amount of vigorous physical activity (h/week) measured using wrist worn accelerometer.
Objective measure of moderate to vigorous physical activity. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The amount of moderate to vigorous physical activity (h/week) measured using wrist worn accelerometer.
Total white matter volume | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Total white matter volumes (mm3) assessed on T1-weighted sequence of brain magnetic resonance imaging.
Total grey matter volume | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Total grey matter volumes (mm3) assessed on T1-weighted sequence of brain magnetic resonance imaging.
Subcortical brain volume of thalamus | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Subcortical brain volume of thalamus (mm3) assessed on T1-weighted sequence of brain magnetic resonance imaging.
Subcortical brain volume of hippocampus | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Subcortical brain volume of hippocampus (mm3) assessed on T1-weighted sequence of brain magnetic resonance imaging.
White matter hyperintensities volume | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Total volume of white matter hyperintensities (mm3) assessed on T2-weighted sequence of brain magnetic resonance imaging.
White matter hyperintensities count | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Total number of white matter hyperintensities on T2-weighted sequence of brain magnetic resonance imaging.
Cerebral vessel lumen diameter | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Cerebral vessel lumen diameter (micrometres) assessed on the time-of-flight sequence of brain magnetic resonance imaging.
Cerebral vessel tortuosity | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The ratio of cerebral vessel tortuosity assessed on the time-of-flight sequence of brain magnetic resonance imaging.
Cerebral vessel density | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Cerebral vessel density (mm3) assessed on the time-of-flight sequence of brain magnetic resonance imaging.
Whole brain grey matter perfusion or cerebral blood flow (CBF) | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Whole brain grey matter perfusion/CBF (in ml/100g/min) assessed on arterial spin labelling of brain magnetic resonance imaging.
Arterial cerebral blood volume fraction | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Arterial cerebral blood volume fraction (%) assessed on arterial spin labelling on brain magnetic resonance imaging.
Circulating vascular endothelial growth factor A as an angiogenic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating vascular endothelial growth factor A (pg/mL) measured from plasma blood samples.
Circulating soluble endoglin as an angiogenic marker. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating soluble endoglin (ng/mL) measured from plasma blood samples.
Circulating soluble fms-like tyrosine kinase-1 as an angiogenic marker. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating soluble fms-like tyrosine kinase-1 measured from plasma blood samples.
Circulating total cholesterol as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of total cholesterol (mmol/L) measured from serum blood samples.
Circulating high-density lipoprotein as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating high-density lipoprotein (mmol/L) measured from serum blood samples.
Circulating low-density lipoprotein as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating low-density lipoprotein (mmol/L) measured from serum blood samples.
Circulating triglycerides as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating triglycerides (mmol/L) measured from serum blood samples.
Circulating fasting glucose concentration as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of fasting glucose (mmol/L) measured from whole blood samples.
Circulating fasting insulin concentration as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of fasting insulin (pmol/L) measured from serum blood samples.
Insulin resistance index as a metabolic marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The index calculated as fasting glucose (mmol/L) x fasting insulin (ulU/mL)/22.5.
Circulating C-reactive protein as an inflammatory marker. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of circulating C-reactive protein (mmol/L) measured from serum blood samples.
Circulating soluble intercellular adhesion molecule-1 (slCAM-1) as an inflammatory marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of sICAM-1 (ng/mL) measured from serum blood samples.
Circulating soluble vascular adhesion molecule-1 (sVCAM-1) as an inflammatory marker | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The level of sVCAM-1 (ng/mL) measured from serum blood samples.
Body weight | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Body weight (kg)
Body height | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Body height (m).
Body mass index (BMI) | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Body weight divided by the square of height (kg/m2).
Mid-arm circumference | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Mid-arm circumference (cm).
Waist-to-hip ratio | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The ratio of waist circumference (cm) to hip circumference (cm).
Systolic blood pressure | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Resting brachial blood pressure measurement (mmHg).
Diastolic blood pressure | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Resting brachial blood pressure measurement (mmHg).
Mean arterial pressure. | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The average arterial pressure from resting brachial blood pressure measurement (mmHg).
Pulse pressure | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The difference between systolic and diastolic blood pressure (mmHg).
Heart rate | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The frequency of the heart contractions per minute (bpm).
Smoking status | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  The number and percentage of current smokers.
Alcohol consumption | Participants will be recruited at 10 to 25 years post index pregnancy and assessed up to 40 years post index pregnancy
  Weekly alcoholic unit intake (units per week).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford Department of Cardiovascular Medicine, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No